CLINICAL TRIAL: NCT06622057
Title: Phase III, Randomized, Double-blind Study of Combination Therapy With D07001-Softgel Capsules and Capecitabine vs Placebo and Capecitabine in Patients With Advanced BTC After Failed on Gemcitabine, Platin, and FOLFOX or Irinotecan Regimens
Brief Title: D07001 Softgel-Capsules and Capecitabine Combination Therapy in Patients With Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InnoPharmax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-GO-07
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer (BTC)
Keywords: BTC; cholangiocarcinoma; Biliary Tract Cancer; third-line
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- D07001-Softgel Capsules 60 mg + Capecitabine (Experimental): * D07001-softgel capsules, 60 mg/day, orally 3 times per week before lunch (on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle)
  * Capecitabine tablets (1000 mg/m2 bid) for 14 days (on Days 1 through 14 of a 21 day cycle) followed by a 7-day rest period. Capecitabine will be taken after breakfast and after dinner.
  Interventions: Drug: D07001-Softgel Capsules; Combination Product: Capecitabine
- D07001-Softgel Capsules 100 mg + Capecitabine (Experimental): * D07001-softgel capsules, 100 mg/day, orally 3 times per week before lunch (on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle)
  * Capecitabine tablets (1000 mg/m2 bid) for 14 days (on Days 1 through 14 of a 21 day cycle) followed by a 7-day rest period. Capecitabine will be taken after breakfast and after dinner.
  Interventions: Drug: D07001-Softgel Capsules; Combination Product: Capecitabine
- Placebo + Capecitabine (Placebo Comparator): * Placebo, orally 3 times per week before lunch (on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle)
  * Capecitabine tablets (1000 mg/m2 bid) for 14 days (on Days 1 through 14 of a 21 day cycle) followed by a 7-day rest period. Capecitabine will be taken after breakfast and after dinner.
  Interventions: Drug: Placebo; Combination Product: Capecitabine

INTERVENTIONS:
Drug: D07001-Softgel Capsules — D07001-softgel capsule is an oral gemcitabine.
  Arms: D07001-Softgel Capsules 100 mg + Capecitabine; D07001-Softgel Capsules 60 mg + Capecitabine
Drug: Placebo — Placebo has the same excipient with D07001-softgel but without active pharmaceutical ingredients (APIs)
  Arms: Placebo + Capecitabine
Combination Product: Capecitabine — Capecitabine, a fluoropyrimidine carbamate derivative, is an oral tumor activator and selective cytotoxic agent.

SUMMARY:
The object of this trial is to evaluate the efficacy of D07001-softgel capsules + capecitabine compared with placebo + capecitabine by overall survival (OS).

Eligible patients with advanced biliary tract cancer (BTC) will be randomized (1:1:1) to receive either 60 mg D07001-softgel, 100 mg D07001-softgel, or placebo, combine with capecitabine. Treatment will be continued until disease progression, death, withdraw consent, or completing 12 treatment cycles , whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, multicenter, placebo-controlled, parallel-group study to evaluate the efficacy and safety of D07001-softgel capsules + capecitabine tablets in participants with advanced BTC after failure on an intravenous gemcitabine and cisplatin-based, and also failed on or refused FOLFOX or failed on irinotecan and fluorouracil regimen. Approximately 195 participants (approximately 65 per treatment arm) will be randomized 1:1:1 to one of the following treatment arms:

* Oral D07001 softgel capsules, 100 mg/day + capecitabine tablets (1000 mg/m2 twice daily [bid])
* Oral D07001 softgel capsules, 60 mg/day + capecitabine tablets (1000 mg/m2 bid)
* Oral placebo softgel capsules + capecitabine tablets (1000 mg/m2 bid) A formal interim futility analysis will be conducted when approximately 80 participants have either experienced disease progression or death. Study participants will continue study treatment until unacceptable toxicity, disease progression, death, withdrawal of consent to treatment, or completing 12 treatment cycles, whichever comes first. The EOT Visit will occur following unacceptable toxicity, disease progression, completing 12 treatment cycles or withdrawal of consent to treatment. Follow-up Period/Visits over phone call will be conducted for participants on 30 ± 3 days, every month; and at 365 ± 3 days following the EOT Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures and agree to adhere to all protocol requirements
2. Aged at least 18 years.
3. Has histopathological or cytologic diagnosis of unresectable, locally advanced or metastatic BTC.
4. Has measurable disease as assessed by RECIST v1.1.
5. Must have failed on a gemcitabine + cisplatin-based chemotherapy, regardless of whether immune checkpoint inhibitor, such as durvalumab or pembrolizumab, or S-1 (tegafur, gimeracil, and oteracil potassium), was also administered. Oxaliplatin or carboplatin may be substituted for cisplatin when renal or auditory function is of concern. Participants also have failed (disease progression or intolerance) on, or refused FOLFOX chemotherapy, including modified FOLFOX variants, or failed on or irinotecan + fluorouracil chemotherapy.
6. Participants with tumors expressing the following biomarkers can be enrolled if they have not previously received FOLFOX but have received appropriate targeted therapies until disease progression or intolerance: fibroblast growth factor receptors aberrations, microsatellite instability biomarker/deficient DNA mismatch repair, or isocitrate dehydrogenase mutations.
7. ECOG PS of 0-2.
8. Life expectancy is ≥12 weeks.
9. Has adequate bone marrow function, demonstrated by: (a) ANC ≥1500 cell/mm3; (b) Platelet count ≥85,000 cells/mm3; (c) Hemoglobin ≥9 g/dL.
10. Has adequate liver function, demonstrated by: (a) AST and ALT ≤2.5 × ULN, or ≤5.0 × ULN in the case of liver lesions; (b) Total bilirubin ≤1.5 × ULN; (c) Albumin ≥3.0 g/dL; (d) INR <1.5.
11. Has adequate renal function, demonstrated by CCR ≥ 45 mL/min or eGFR ≥ 45 mL/min/1.73 m2
12. No clinically significant abnormalities in coagulation results.
13. Participant is eligible to participate if not pregnant (as demonstrated by serum pregnancy testing at screening), not breastfeeding, and at least 1 of the following conditions applies:

    1. Not of childbearing potential (CBP).
    2. A participant of CBP who is sexually active with a partner who could impregnate them agrees to use a highly effective form of contraception during the study and for at least 30 days after the end of study intervention.
14. With partners of childbearing potential whom they could impregnate must agree to use contraception during the study and for 90 days after the end of study intervention.
15. Participants who are able to donate sperm must refrain from sperm donation during the study and for 90 days after the end of study intervention.
16. Participant is willing to comply with the protocol-required visit schedule and visit requirements.
17. More than 14 days have elapsed between the participant completing a prior line of chemotherapy or target therapy, and enrollment. More than 28 days have elapsed between the participant receiving concurrent radiotherapy (CCRT) and enrollment.

Exclusion Criteria:

1. Has a diagnosis of active malignancy other than BTC within the past 2 years, except nonmelanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent.
2. Participant discontinued prior gemcitabine due to pulmonary or hepatic toxicity or hemolytic uremic syndrome, hypersensitivity, allergic reaction, or intolerance.
3. Participant had a prior unanticipated severe reaction to capecitabine or metabolites or to fluoropyrimidine therapy.
4. Participant received treatment with brivudine, sorivudine, or its chemically related analogs ≤28 days prior to the date of enrollment.
5. Participant is currently receiving flucytosine treatment.
6. Participant has residual toxicity from prior chemotherapy or CCRT that is Grade ≥2 (residual Grade 2 neuropathy and alopecia are permitted).
7. Participant has any gastrointestinal disorder or prior gastrointestinal surgery that would significantly impede absorption of an oral agent, such as gastrectomy, Crohn's disease, ulcerative colitis, or short gut syndrome.
8. Participant has known brain or leptomeningeal metastases.
9. Participant had major surgery or definitive ablation-intent (excluding palliative radiotherapy for bone metastasis) radiation therapy within the past 28 days.
10. Participant has any active disease or condition that would not permit compliance with the protocol.
11. Participant has clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, congestive heart failure, New York Heart Association Grade 2 or greater), or uncontrolled serious cardiac arrhythmia.
12. Participant has documented cerebrovascular disease.
13. Participant has a seizure disorder not controlled with medication (based on Investigator's decision).
14. Participant has received an investigational agent within 28 days of enrollment.
15. Participant has an uncontrolled active viral, bacterial, or systemic fungal infection.
16. Participant has positive hepatitis B surface antigen with positive hepatitis B virus DNA ≥2000 copies/mL and/or anti-hepatitis C virus antibody.
17. Participant has received yellow fever vaccine or other live attenuated vaccine(s) within the 4 weeks before screening.
18. Participant has a history of drug or alcohol abuse within the year before signing the informed consent form.
19. Participant has any other serious medical condition that, in the Investigator's medical opinion, would preclude safe participation in or compliance with the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death, assessed up to 2 years
  To assess the over survival (OS) of 2 doses of D07001-softgel capsules + capecitabine compared with placebo + capecitabine

SECONDARY OUTCOMES:
progression-free survival (PFS) | From randomization to death or progression disease, assessed up to 2 years
  To assess the progression-free survival (PFS) of D07001-softgel capsules + capecitabine compared with placebo + capecitabine
6-month survival rate | Assessed as the time at 6 month timepoint from randomization
  To assess the 6-month OS of D07001-softgel capsules + capecitabine compared with placebo + capecitabine
overall response rate (ORR) | From treatment starting until end of treatment(EOT), assessed up to complete 12 treatment cycles (each cycle is 21 days).
  To assess the overall response rate (ORR) of D07001-softgel capsules + capecitabine
Quality of life (QOL) will be assessed using the EORTC questionnaires | Assessed as the time from randomization to end of treatment(EOT), assessed up to complete 12 treatment cycles (each cycle is 21 days).
  To access healthy related quality of life of cancer patients participating in clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Huang, Study Director — InnoPharmax Inc.
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No